CLINICAL TRIAL: NCT05937308
Title: Interventional Registry to Collect Real-World Evidence of the NEUROMARK System in Subjects With Chronic Rhinitis
Brief Title: NEUROMARK Registry Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neurent Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-0008
Record Dates: First submitted 2023-06-16; First posted 2023-07-10 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-09

CONDITIONS: Chronic Rhinitis
Keywords: Rhinitis
MeSH Terms: conditions — Rhinitis

STUDY DESIGN:
Intervention Model Description: A Prospective, Multicenter, Single-arm, Post-market Interventional Registry. Collect real-world evidence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- NEUROMARK Treatment (Other): Interventional registry to collect real world data - Subjects will undergo treatment with the NEUROMARK System.
  Interventions: Device: NEUROMARK System

INTERVENTIONS:
Device: NEUROMARK System — The NEUROMARK System is indicated for use in otorhinolaryngology (ENT) surgery for creation of radiofrequency (RF) lesions to disrupt posterior nasal nerves in patients with chronic rhinitis.

SUMMARY:
The NEUROMARK Registry Study is a prospective, multicenter, single-arm, post-market, interventional registry study to collect real-world evidence of the NEUROMARK System in subjects with chronic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

Subject MUST:

1. Be ≥18 years of age.
2. Be scheduled to receive treatment with the commercially available NEUROMARK System consistent with the device's indications for use.
3. Have moderate to severe symptoms of running nose (individual rTNSS symptom rating of 2 or 3), mild to severe symptoms of nasal congestion (individual rTNSS symptom rating of 1, 2, or 3), and a minimum total score of 5 (out of 12) at screening.
4. Be willing and able to provide consent and comply with all study elements, as indicated by written informed consent.

Exclusion Criteria:

Subjects Must Not:

1. Have a history of chronic epistaxis or experienced a significant epistaxis event (defined as epistaxis requiring medical intervention) in the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Safety - incidence of device- and/or procedure-related serious adverse | 3-month follow-up
  Safety, as assessed by the incidence of device- and/or procedure-related serious adverse events (SAEs).
Safety - incidence of device- and/or procedure-related serious adverse | 6-month follow-up
  Safety, as assessed by the incidence of device- and/or procedure-related serious adverse events (SAEs).
Safety - incidence of device- and/or procedure-related serious adverse | 12-month follow-up
  Safety, as assessed by the incidence of device- and/or procedure-related serious adverse events (SAEs).
Safety - incidence of device- and/or procedure-related serious adverse | 18-month follow-up
  Safety, as assessed by the incidence of device- and/or procedure-related serious adverse events (SAEs).
Safety - incidence of device- and/or procedure-related serious adverse | 24-month follow-up
  Safety, as assessed by the incidence of device- and/or procedure-related serious adverse events (SAEs).
Safety - incidence of device- and/or procedure-related serious adverse | 30-month follow-up
  Safety, as assessed by the incidence of device- and/or procedure-related serious adverse events (SAEs).
Safety - incidence of device- and/or procedure-related serious adverse | 36-month follow-up
  Safety, as assessed by the incidence of device- and/or procedure-related serious adverse events (SAEs).
Efficacy - reflective Total Nasal Symptom Score (rTNSS) | 3-month follow-up
  Efficacy, as assessed by the mean change from baseline in the reflective Total Nasal Symptom Score (rTNSS) total score at each follow-up
Efficacy - reflective Total Nasal Symptom Score (rTNSS) | 6-month follow-up
  Efficacy, as assessed by the mean change from baseline in the reflective Total Nasal Symptom Score (rTNSS) total score at each follow-up
Efficacy - reflective Total Nasal Symptom Score (rTNSS) | 12-month follow-up
  Efficacy, as assessed by the mean change from baseline in the reflective Total Nasal Symptom Score (rTNSS) total score at each follow-up
Efficacy - reflective Total Nasal Symptom Score (rTNSS) | 18-month follow-up
  Efficacy, as assessed by the mean change from baseline in the reflective Total Nasal Symptom Score (rTNSS) total score at each follow-up
Efficacy - reflective Total Nasal Symptom Score (rTNSS) | 24-month follow-up
  Efficacy, as assessed by the mean change from baseline in the reflective Total Nasal Symptom Score (rTNSS) total score at each follow-up
Efficacy - reflective Total Nasal Symptom Score (rTNSS) | 30-month follow-up
  Efficacy, as assessed by the mean change from baseline in the reflective Total Nasal Symptom Score (rTNSS) total score at each follow-up
Efficacy - reflective Total Nasal Symptom Score (rTNSS) | 36-month follow-up
  Efficacy, as assessed by the mean change from baseline in the reflective Total Nasal Symptom Score (rTNSS) total score at each follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Annalise Sorensen, Study Director — Neurent Medical
Locations (7):
- United States (7):
  - Alabama Nasal & Sinus Center, Birmingham, Alabama
  - Sensa Health, Los Angeles, California
  - Sacramento ENT, Roseville, California
  - Florida ENT & Allergy, Brandon, Florida
  - ENT & Allergy Texas, McKinney, Texas
  - Ogden Clinic, Ogden, Utah
  - Metropolitan ENT, Alexandria, Virginia

IPD SHARING:
Plan to Share IPD: No